CLINICAL TRIAL: NCT01936155
Title: Does Neuromuscular Electrical Stimulation (NMES) Help Relieve Lower Limb Oedema and Improve Joint Mobility and Skin Tissue Oxygenation Levels?
Brief Title: Does NMES Help Relieve Lower Limb Oedema and Improve Joint Mobility and Skin Tissue Oxygenation Levels?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Merlin Park University Hospital, Galway, Ireland (Unknown)
Responsible Party: Principal Investigator, Gearoid O Laighin, Professor, National University of Ireland, Galway, Ireland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EE-NMES-OED-336
Record Dates: First submitted 2013-09-02; First posted 2013-09-05 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Oedema
Keywords: Joint Mobility; Skin Tissue Oxygenation; Neuromuscular Electrical Stimulation; Goniometry; Transcutaneous Oxygen Measurements (tcpO2); Water Displacement
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oedema, Joint Mobility, Skin Oxygenation (Experimental): Neuromuscular electrical stimulation (NMES) is to be applied using a custom-built, two-channel stimulator, Bioelectronics Research Cluster, National University of Ireland, Galway) with a frequency of 36 Hz, a balanced biphasic waveform with a pulse width of 350μs, a ramp up time of 500ms, a contraction time of 1s and a ramp down time of 500ms. Stimulation is to be applied every 20 seconds over a period of 90 minutes. Its affect on oedema reduction, joint mobility and skin oxygenation will be assessed both before and after its application.
  Interventions: Device: Custom-built, two-channel stimulator

INTERVENTIONS:
Device: Custom-built, two-channel stimulator — Custom-built, two-channel stimulator for stimulation of the soleus calf muscle

SUMMARY:
Neuromuscular Electrical Stimulation (NMES) will be facilitated through the use of a stimulator, with the patient in a semi recumbent position, using UltraStim electrodes. Two 5 cm x 5 cm electrodes will be placed over the soleus muscle for calf stimulation. The participant will be allowed to ramp up the stimulus level themselves to get used to the sensation and determine their maximum tolerated stimulus level.

A goniometer will be used to assess mobility at the knee and ankle joints. Transcutaneous oxygen measurements (tcpO2) will be assessed using the PERIMED Periflux System 500 tcpO2 monitor.

The level of oedema will be measured using the figure of eight measurement, tape circumference measurement and water displacement measurement.

Comfort will also be assessed by use of a 100mm non-hatched visual analogue scale (VAS). Each participant will be asked to indicate their level of comfort following the application of NMES.

DETAILED DESCRIPTION:
Neuromuscular Electrical Stimulation (NMES) will be facilitated through the use of a two-channel, research stimulator, with the patient in a semi recumbent position, using UltraStim electrodes. Two 5 cm x 5 cm electrodes will be placed over the soleus muscle for calf stimulation. The participant will be allowed to ramp up the stimulus level themselves to get used to the sensation and determine their maximum tolerated stimulus level.

A goniometer will be used to assess mobility at the knee and ankle joints. Transcutaneous oxygen measurements (tcpO2) will be assessed using the PERIMED Periflux System 500 tcpO2 monitor.

The level of oedema will be measured using the figure of eight measurement, tape circumference measurement and water displacement measurement.

Comfort will also be assessed by use of a 100mm non-hatched visual analogue scale (VAS). Each participant will be asked to indicate their level of comfort following the application of NMES. VAS pain scores of 30 mm or less will be categorised as mild pain, between 31 and 69 mm as moderate pain, and scores of 70 mm or greater as severe pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients that present to Merlin Park Podiatry Clinic for Podiatric Intervention who on clinical examination present with lower lib swelling/oedema/
* Ability to understand the nature of the study.
* Ability to give informed consent.

Exclusion Criteria:

* Skin ulceration in area of intended electrical stimulation site.
* Psychiatric disorder.
* Severe co-morbidity.
* Patients with uncontrolled heart problems.
* Patients with pacemakers, DBS.
* Patients on opioid or neuropathic pain medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Oedema Reduction | Approximately three and a half hours
  Oedema measurements (figure of eight measurement, tape circumference measurement and water displacement measurement) will be taken before and after the application of neuromuscular electrical stimulation (NMES) in order to assess its affect on the reduction of oedema.

SECONDARY OUTCOMES:
Joint Mobility | Approximately three and a half hours
  A goniometer will be used to assess mobility at the ankle and knee joints both before and after the application of neuromuscular electrical stimulation (NMES) to the soleus muscle of the calf.
Skin Oxygenation | Approximately three and a half hours
  Transcutaneous oxygen measurements (tcpO2) will be assessed using the PERIMED Periflux System 5000 tcpO2 monitor both before and after the application of NMES to the soleus muscle in order to assess its affect on skin tissue oxygenation levels.

CONTACTS AND LOCATIONS:
Overall Officials: David Watterson, BSc Podiatry, Principal Investigator — Merlin Park University Hospital, Galway, Ireland
Locations (1):
- Merlin Park University Hospital, Galway, Ireland